CLINICAL TRIAL: NCT01368276
Title: An Extension Protocol to Evaluate the Efficacy and Safety of Extended Use Treatment With OncoVEX^GM-CSF for Eligible Melanoma Patients Participating in Study 005/05
Brief Title: An Extended Use Study of Safety and Efficacy of Talimogene Laherparepvec in Melanoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioVex Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 005/05-E; 2010-021070-11 (EudraCT Number); 20110279 (Other: Sponsor)
Record Dates: First submitted 2011-04-20; First posted 2011-06-07 (Estimated); Results first posted 2015-12-18 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-11

CONDITIONS: Melanoma
Keywords: Melanoma; Stage IIIb, IIIc and IV Disease; oncolytic; OncoVex; OncoVEX^GM-CSF
MeSH Terms: conditions — Melanoma | interventions — talimogene laherparepvec; Colony-Stimulating Factors; Granulocyte-Macrophage Colony-Stimulating Factor

ARMS (2):
- GM-CSF (Active Comparator): Granulocyte macrophage colony-stimulating factor (GM-CSF) was administered at a dose of 125 μg/m²/day subcutaneously for 14 consecutive days followed by 14 days of rest, in 28-day treatment cycles for up to 12 months or until a complete response, occurrence of an unacceptable toxicity, death or another criterion for withdrawal from treatment was met. Participants who demonstrated a partial response after being on treatment for 12 months could continue to be treated until disease progression or another treatment discontinuation criterion was met.
  Interventions: Drug: Granulocyte Macrophage Colony-Stimulating Factor (GM-CSF)
- Talimogene Laherparepvec (Experimental): Talimogene laherparepvec was administered at a concentration of 10⁸ plaque forming units (PFU)/mL injected into 1 or more skin or subcutaneous tumors on Days 1 and 15 of each 28-day cycle for up to 12 months or until a complete response, occurrence of an unacceptable toxicity, death or another criterion for withdrawal from treatment was met. Participants who demonstrated a partial response after being on treatment for 12 months could continue to be treated until disease progression or another treatment discontinuation criterion was met.
  Interventions: Biological: Talimogene Laherparepvec

INTERVENTIONS:
Biological: Talimogene Laherparepvec — Up to 4 mL of 10⁸ pfu/mL/per intratumoral injection
  Other Names: OncoVEX^GM-CSF; IMLYGIC™
  Arms: Talimogene Laherparepvec
Drug: Granulocyte Macrophage Colony-Stimulating Factor (GM-CSF) — 125 µg/m² subcutaneous injection
  Arms: GM-CSF

SUMMARY:
The purpose of this study is to learn about the safety and the risks of using talimogene laherparepvec in patients who already received treatment with talimogene laherparepvec in study 005/05 (NCT00769704), and to see if extended treatment with talimogene laherparepvec can destroy melanoma tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Previously participated in protocol 005/05 (NCT00769704) and:

   1. received the maximum number of talimogene laherparepvec treatment injections or cycles of GM-CSF allowable for that patient on study 005/05, or
   2. new injectable lesion(s) appeared after previous resolution of all injectable disease while on study 005/05. New injectable lesions must have appeared within ≤ 12 months from the End of Treatment visit on the 005/05 study.
2. In the opinion of the investigator and the sponsor's medical monitor further treatment is warranted [e.g., those patients who do not have clinically relevant progressive disease (PDr)].
3. Performance status (Eastern Cooperative Oncology Group, ECOG) 0 or 1.
4. For patients randomized to talimogene laherparepvec only: Injectable disease (i.e. suitable for direct injection or through the use of ultrasound guidance) defined as at least 1 injectable cutaneous, subcutaneous or nodal melanoma lesion. There is no minimum size for injection.

Exclusion Criteria:

1. Prior Common Terminology Criteria for Adverse Events (CTCAE) grade 3 or 4 toxicity related to talimogene laherparepvec of any organ system (with the exception of injection site reactions, fever and vomiting).
2. History of Grade 3 fatigue lasting > 1 week while on talimogene laherparepvec treatment.
3. History of Grade 3 arthralgia/myalgias while on talimogene laherparepvec treatment.
4. History of ≥ Grade 2 autoimmune reactions, allergic reactions or urticaria or other talimogene laherparepvec related non-hematological toxicities while on talimogene laherparepvec treatment that required a dose delay or discontinuation of talimogene laherparepvec therapy.
5. PDr while participating in study 005/05
6. Patient requested to be withdrawn from study 005/05 or was unable to comply with the demands of the 005/05 trial.
7. At the discretion of the investigator, patient was withdrawn from the 005/05 trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (9):
  - Rush University Medical Center, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Hubert H Humphrey Cancer Center, Robbinsdale, Minnesota
  - University of North Carolina At Chapel Hill School of Medicine, Chapel Hill, North Carolina
  - Mary Crowley Medical Research Center, Dallas, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Oncology and Hematology Associates of Southwest Virginia, Inc., Salem, Virginia
- Royal Marsden Hospital, London, United Kingdom

REFERENCES:
- See also: Sponsor Website — http://www.biovex.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This extension was available to patients who participated in study 005/05 (NCT00769704), received the maximum allowable number of treatments or developed new lesion(s) within ≤ 12 months from the end of treatment visit after previous resolution of all disease while on study 005/05, and warranted further treatment per the investigator.
Pre-assignment Details: Participants received the same treatment as randomized under the 005/05 study.
Period: Overall Study
Arm/Group | GM-CSF | Talimogene Laherparepvec
Started | 3 | 28
Completed | 2 | 18
Not Completed | 1 | 10
Not completed — Death | 1 | 10

BASELINE CHARACTERISTICS:
Groups:
- GM-CSF: GM-CSF was administered at a dose of 125 μg/m²/day subcutaneously for 14 consecutive days followed by 14 days of rest, in 28-day treatment cycles for up to 12 months or until a complete response, occurrence of an unacceptable toxicity, death or another criterion for withdrawal from treatment was met. Participants who demonstrated a partial response after being on treatment for 12 months could continue to be treated until disease progression or another treatment discontinuation criterion was met.
- Talimogene Laherparepvec: Talimogene laherparepvec was administered at a concentration of 10⁸ PFU/mL injected into 1 or more skin or subcutaneous tumors on Days 1 and 15 of each 28-day cycle for up to 12 months or until a complete response, occurrence of an unacceptable toxicity, death or another criterion for withdrawal from treatment was met. Participants who demonstrated a partial response after being on treatment for 12 months could continue to be treated until disease progression or another treatment discontinuation criterion was met.
- Total: Total of all reporting groups
Arm/Group | GM-CSF | Talimogene Laherparepvec | Total
Number analyzed (Participants) | 3 | 28 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (25.0) | 64.2 (13.2) | 63.3 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 14 | 16
  Male | 1 | 14 | 15
Race/Ethnicity, Customized [Number; unit: participants]
  White | 3 | 28 | 31
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Scale used to assess how a patient's disease is progressing, how the disease affects the daily living abilities of the patient: 0 = Fully active, able to carry on all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity, ambulatory, able to carry out work of a light nature; 2 = Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about > 50% of waking hours; 3 = Capable of only limited self care, confined to a bed or chair > 50% of waking hours; 4 = Completely disabled, confined to bed or chair; 5 = Dead.
  participants
    0 | 3 | 20 | 23
    1 | 0 | 8 | 8
Disease Stage [Number; unit: participants] — Stage IIIB: Ulcerated lesion and 1 lymph node or 2-3 nodes with micrometastasis, or any-depth lesion with no ulceration, and 1 lymph node or 2-3 nodes with macrometastasis; Stage IIIC: Ulcerated lesion and 1 lymph node with macrometastasis; 2-3 nodes with macrometastasis or ≥ 4 metastatic lymph nodes, matted lymph nodes, or in-transit met(s)/satellite(s); Stage IV: M1a: Spread to skin, subcutaneous tissue, or lymph nodes; normal lactate dehydrogenase (LDH) level; M1b: Spread to lungs; normal LDH; M1c: Spread to all other visceral organs, normal LDH or any distant disease with elevated LDH.
  participants
    Stage IIIB | 0 | 1 | 1
    Stage IIIC | 0 | 6 | 6
    Stage IV M1a | 1 | 9 | 10
    Stage IV M1b | 1 | 8 | 9
    Stage IV M1c | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (AEs)
Description: AEs were graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 3.0 based on the following guideline:
  Grade 1: Mild AE; Grade 2: Moderate AE; Grade 3: Severe AE; Grade 4: Life-threatening or disabling AE; Grade 5: Death related to AE.
  Treatment-related AE refers to AEs that have possible or probable relation to study treatment as determined by the investigator.
  A serious AE is one that meets one or more of the following criteria/outcomes:
  * Results in death.
  * Is life-threatening.
  * Requires inpatient hospitalization or prolongation of existing hospitalization.
  * Results in persistent or significant disability/incapacity.
  * Is a congenital anomaly/birth defect.
  * Is an important medical event.
Time Frame: From first administration of study drug in the extension period until 30 days after last dose. Median duration of treatment was 50 weeks in the GM-CSF group and 36 weeks in the talimogene laherparepvec group.
Population: Safety population (randomized participants who received at least one dose of extension treatment).
Measure: Number; unit: participants
Arm/Group | GM-CSF | Talimogene Laherparepvec
Number analyzed (Participants) | 3 | 28
participants
  All adverse events | 3 | 26
  Worst grade of 3 | 0 | 5
  Worst grade of 4 | 0 | 1
  Worst grade of 5 | 0 | 2
  Serious adverse events | 0 | 9
  Treatment-related adverse events | 3 | 20
  Treatment-related serious adverse events | 0 | 1
  Leading to discontinuation of study treatment | 0 | 4
  Leading to study treatment delay | 0 | 4
  Fatal adverse events on-study | 0 | 2

2. Secondary Outcome: Objective Response Rate
Description: Objective response rate was defined as the percentage of participants with a best overall response of complete response (CR) or partial response (PR) assessed by the investigator. Best overall response for a patient is the best overall response observed across all time points and is cumulative (ie, includes responses during the parent study 005/05 and during Study 005/05-E).
  Disease assessments were performed at the beginning of each treatment cycle and assessed in accordance with modified World Health Organization criteria.
  CR: Disappearance of all clinical evidence of tumor (both measurable and non-measurable but evaluable disease); PR: ≥ 50% reduction in the sum of the products of the perpendicular diameters of all measurable tumors at the time of assessment as compared to baseline.
Time Frame: From randomization in study 005/05 until the data-cut-off date for the extension period of 08 August 2014; median treatment duration for 005/05 and 005/05-E studies combined was 88 weeks for talimogene laherparepvec and 100 weeks for GM-CSF.
Population: The full analysis set for the extension study is defined as all participants who received at least one dose of extension treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GM-CSF | Talimogene Laherparepvec
Number analyzed (Participants) | 3 | 28
percentage of participants | 100.0 [NA to NA] — For 100% response, the asymptotic 95% CI was not estimated since the mathematical formula is not considered appropriate in such extreme cases. | 57.1 [38.8 to 75.5]
Statistical Analysis 1: Comparison: GM-CSF vs Talimogene Laherparepvec; Test type: Superiority or Other; p = 0.2645, Fisher Exact — Descriptive; Treatment Difference = -42.9 — Talimogene laherparepvec - GM-CSF

3. Secondary Outcome: Durable Response Rate
Description: Durable response rate is defined as the percentage of participants with a complete response (CR) or partial response (PR) assessed by the investigator, initiating at any time while receiving talimogene laherparepvec or GM-CSF therapy on the 005/05 or the 005/05-E study and maintained continuously for at least 6 months from response initiation. This reflects all new sites of disease as well as disease sites identified at baseline.
  Disease assessments were performed at the beginning of each treatment cycle in accordance with modified World Health Organization criteria.
  CR: Disappearance of all clinical evidence of tumor (both measurable and non-measurable but evaluable disease); PR: ≥ 50% reduction in the sum of the products of the perpendicular diameters of all measurable tumors at the time of assessment as compared to baseline.
Time Frame: as for outcome 2
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GM-CSF | Talimogene Laherparepvec
Number analyzed (Participants) | 3 | 28
percentage of participants | 33.3 [0.0 to 86.7] | 32.1 [14.8 to 49.4]
Statistical Analysis 1: Comparison: GM-CSF vs Talimogene Laherparepvec; Test type: Superiority or Other; p = 1.0000, Fisher Exact — Descriptive; Treatment Difference = -1.2, 95% CI 2-sided [-57.3 to 54.9] — Talimogene laherparepvec - GM-CSF

ADVERSE EVENTS:
Time Frame: From first administration of study drug in the extension period until 30 days after last dose. Median duration of treatment was 50 weeks in the GM-CSF group and 36 weeks in the talimogene laherparepvec group.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | GM-CSF | Talimogene Laherparepvec
Serious Adverse Events (participants affected / at risk) | 0/3 | 9/28
Other Adverse Events (participants affected / at risk) | 3/3 | 21/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GM-CSF (N=3) | Talimogene Laherparepvec (N=28)
Cardiac arrest (Cardiac disorders) | 0 | 1
Restrictive cardiomyopathy (Cardiac disorders) | 0 | 1
Disease progression (General disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 1
Vasculitis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GM-CSF (N=3) | Talimogene Laherparepvec (N=28)
Ear pain (Ear and labyrinth disorders) | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 4
Nausea (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 1 | 3
Chills (General disorders) | 1 | 5
Fatigue (General disorders) | 2 | 3
Influenza like illness (General disorders) | 1 | 1
Injection site mass (General disorders) | 1 | 0
Injection site pain (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 1 | 3
Pyrexia (General disorders) | 1 | 5
Folliculitis (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Dizziness (Nervous system disorders) | 0 | 3
Headache (Nervous system disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypopnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Blood blister (Skin and subcutaneous tissue disorders) | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 3
Flushing (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.